CLINICAL TRIAL: NCT03853187
Title: Imaging Tumor-infiltrating CD8+ T-cells in Non-small Cell Lung Cancer Upon Neo-adjuvant Treatment With Durvalumab (MEDI4736)
Brief Title: Imaging Tumor-infiltrating T-cells in Non-small Cell Lung Cancer
Acronym: Donan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-17-13332; NL68987.091.19 (Registry Identifier: Dutch trial registry); 2019-000670-37 (EudraCT Number)
Record Dates: First submitted 2019-02-11; First posted 2019-02-25 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (MEDI4736) neo-adjuvant (Experimental): Patients will receive two courses of durvalumab (MEDI4736)at a fixed dose of 750mg Q2W intravenously, prior to scheduled resection of NSCLC. Patients are amendable to adjuvant chemo and/or radiation treatment, per standard-of-care. Additionally, patients will undergo a Zr-89 labelled durvalumab (MEDI4736) PET/CT and dedicated perfusion-CT prior to treatment with durvalumab (MEDI4736) and ex vivo In-111-oxine or in vivo [89Zr]-Df-crefmirlimab labelled CD8+ T-cells after two courses of treatment, prior to surgery.
  Interventions: Radiation: Zr-89 labelled durvalumab PET/CT; Drug: Durvalumab (MEDI4736)

INTERVENTIONS:
Radiation: Zr-89 labelled durvalumab PET/CT — Patients will undergo a Zr-89 labelled durvalumab (MEDI4736) PET/CT and dedicated perfusion-CT prior to treatment with durvalumab (MEDI4736) and in- and ex-vivo In-111-oxine or in-vivo [89zr]-Df-crefmirlimab labelled CD8+ T-cells after two courses of treatment, prior to surgery.
  Other Names: In-111-oxine labelled CD8+ T-cell scintigraphy OR [89Zr]-Df-crefmirlimab PET; Dedicated perfusion-CT
Drug: Durvalumab (MEDI4736) — Patients will receive two courses of durvalumab (MEDI4736)at a fixed dose of 750mg Q2W intravenously, prior to scheduled resection of NSCLC.

SUMMARY:
This is an interventional study, to assess feasibility and safety of durvalumab (MEDI4736) in neo-adjuvant setting in patients with resectable NSCLC. Additional analyses of potential imaging biomarkers, e.g. Zr-89 labelled durvalumab (MEDI4736), ex vivo In-111-oxine labelled CD8+ T-cells and high-resolution immune cell imaging, in relation to immunotherapy induced immune responses on quantitative immune histochemical analysis of the resected tumor specimen, will be performed.

DETAILED DESCRIPTION:
This is an interventional study in 20 patients with resectable non-small cell lung cancer who will receive 2 courses of durvalumab (MEDI4736) in the neo-adjuvant setting, followed by surgery with curative intent.

Experimental imaging procedures include 1) Zr-89-labelled durvalumab (MEDI4736) scan prior to neo-adjuvant treatment to determine accessibility and intra-tumoral distribution of durvalumab (MEDI4736) and 2) (first cohort) injection of ex vivo [111In]-oxine labelled autologous CD8+ T-cells 48 hours prior to surgery, or (second cohort) injection of [89Zr]-Df-crefmirlimab prior to surgery. The scan is scheduled on the day of surgery and after surgery, the resected tumor specimen with ex vivo [111In]-oxine labelled or in vivo [89Zr]-Df-crefmirlimab labelled CD8+ T-cells in situ, is fixated for high-resolution ex vivo imaging on a preclinical U-SPECT scanner and quantitative histopathological analysis, next to standard histopathological evaluation.

Total duration of the study is maximum 42 days (from injection therapeutic dose durvalumab (MEDI4736) to surgery).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >50 years at time of study entry
* Histopathological proven primary non-small cell lung cancer, with fully evaluable histological biopsies available
* ECOG performance status of 0 or 1
* AJCC stage I, II or IIIa as determined by contrast-enhanced CT chest-abdomen and F-18-FDG PET/CT: cT1cN0-1M0, cT2aN0-1M0 en cT3N0-1M0 (T3 separate nodule)
* Solid appearance of the tumor on contrast-enhanced CT
* Scheduled for resection with curative intent
* Patients should be medically operable defined by:
* Sufficient cardiopulmonary function
* Major contra-indications for surgery.
* No underlying immune disease (neutro- or lymphopenia, coagulation disorders) that could interfere with T-cell isolation
* Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g, Health Insurance Portability and Accountability Act in the US, European Union Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Must have a life expectancy of at least 6 months
* Adequate normal organ and marrow function as defined below:

  * Haemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) 1.5x (> 1500 per ml)
  * Platelet count ≥100 x10^9/L (>75,000 per ml)
* Serum bilirubin ≤1.5x upper limit of normal (ULN). Note: This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST/ALT ≤2.5x upper limit of normal
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (CCL):
* Males: CCL (mL/min) = (Weight (kg) x (140 - Age)) / 72 x serum creatinine (mg/dL)
* Females: CCL (mL/min) = (Weight (kg) x (140 - Age)) / 72 x serum creatinine (mg/dL), multiplied by correction factor 0.85
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Highly effective contraception for both male and female subjects throughout the study and for at least after durvalumab (MEDI4736) treatment administration intrinsic factor the risk of conception exists

Exclusion Criteria:

* Inability to lie supine for more than 30 minutes
* Documented previous severe allergic reaction to iodine-based contrast media, despite adequate pre-medication. In case of documented mild to moderate allergic reaction to iodine-based contrast media, patients will receive premedication according to the local protocol, consisting of 25mg prednisolone intravenously 30 minutes prior to iodine-based contrast media administration and 2mg clemastine intravenously just prior to administration.
* Indication for cervical mediastinoscopy according to the local multidisciplinary Thoracic-Oncology meeting
* Participation in another clinical study with an investigational product during the past 6 months
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) <6 months prior to the first dose of study drug
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab (MEDI4736) may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 6 months of the first dose of study drug
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
  * Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of active primary immunodeficiency
* Active infection including:

  * tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice),
  * hepatitis B (known positive HBV surface antigen (HBsAg) result),
  * hepatitis C,
  * human immunodeficiency virus (positive HIV 1/2 antibodies),
  * Epstein Barr Virus (EBV, positive IgM antibodies)
  * cytomegalo virus (CMV, positive IgM antibodies) NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab (MEDI4736). The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions, e.g. CT scan
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab (MEDI4736). Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab (MEDI4736) and up to 30 days after the last dose of durvalumab (MEDI4736).
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab (MEDI4736) monotherapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Safety of neo-adjuvant durvalumab: number of NCI CTCAE v 5.0 grade ≥3 | 14 days
  Demonstrate safety of two courses durvalumab (MEDI4736) 750 mg at two weeks interval in neo-adjuvant setting. Safety is defined as the number of NCI CTCAE v 5.0 grade ≥3 toxicity related to neo-adjuvant durvalumab (MEDI4736).
Feasibility of neo-adjuvant durvalumab: successful completion of curative surgery | 42 days
  Demonstrate feasibility of two courses durvalumab (MEDI4736) 750 mg at two weeks interval in neo-adjuvant setting. Feasibility is defined as successful completion of curative surgery within 42 days after start of neo-adjuvant treatment with durvalumab (MEDI4736) (= day 1).

SECONDARY OUTCOMES:
Imaging related_response on CE-CT | 42 days
  Objective responses measured on contrast enhanced CT (RECIST1.1, immune related response criteria (irRC))
Imaging related_pathological response | 42 days
  The rate of (major and complete) pathological responses as previously defined.
Imaging related_correlation with Zr89-labelled durvalumab | 42 days
  Correlate the presence and localisation of TILs with the intra-tumoral distribution of Zr-89-labelled durvalumab (MEDI4736).
Imaging related_correlation with perfusion-CT | 42 days
  Correlate the presence and localisation of TILs and Zr-89-labelled durvalumab (MEDI4736) with (changes in) perfusion parameters on contrast-enhanced CT.
Biomarker related_future correlation with other biomarkers | 42 days
  Exploration of In-111-oxine or [89Zr]-Df-crefmirlimab labelled T-cells U-SPECT or PET findings with other potential biomarkers (not yet defined) for response to immune therapy and the number of immune therapy related conversions from VATS to open surgical procedures
Biomarker related_correlation with immune profiling | 42 days
  Correlate the presence of TILs with multi-dimensional immune profiling by flow cytometry of freshly isolated peripheral blood lymphocytes.
Clinical care related_evaluation of VATS conversions | 42 days
  Evaluate the number of VATS conversions after neo-adjuvant durvalumab (MEDI4736).
Clinical care related_number of patients with postoperative complications | 42 days
  Asses postoperative complications
Clinical care related_hospital stay | 42 days
  Asses length of hospital stay
Clinical care related_mortality | 30 and 90 days
  Asses 30 and 90 day mortality
Clinical care related_evaluation of patient related outcomes | 42 days
  Patient related outcome measurements (PROMS) will be evaluated based on the EORTC-QLQ-C30 (quality of life) questionnaire (in Dutch) at baseline, prior to surgery, at first post-operative visit and follow-up.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Clinical care related_determination of recurrence-free survival | 42 days
  Determine recurrence-free survival by landmarking analysis, based on time since surgery.
Clinical care related_determination of overall survival | 42 days
  Determine overall survival by landmarking analysis, based on time since surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Aarntzen, MD, PhD, Principal Investigator — Radboud University Medical Center; Michel van den Heuvel, MD, PhD, Principal Investigator — Radboud University Medical Center; Jolanda de Vries, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No